CLINICAL TRIAL: NCT00820196
Title: A Randomized, Double-Blind, Vehicle-controlled, Parallel Group, Dose-Ranging, Multi-center Study of the Efficacy and Safety of Nexagon® in the Treatment of Participants With Venous Leg Ulcers
Brief Title: A Trial to Assess the Safety and Activity of Nexagon® for the Treatment of Venous Leg Ulcers (The NOVEL Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OcuNexus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEX-ULC-001
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Venous Ulcer
Keywords: Venous ulcer; Nexagon; CoDa
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nexagon®
Drug: Nexagon® vehicle

SUMMARY:
Venous leg ulcers are a common, costly and debilitating condition, with few effective treatments. Compression bandaging helps healing, but more than four out of every ten leg ulcers remain unhealed after three months. New treatments to help heal venous ulcers are urgently needed. Initial studies with a new drug product candidate called Nexagon® (developed by CoDa Therapeutics, Inc.) have shown improvements in healing when applied topically to a wound. Further research will be undertaken to assess the safety and activity of Nexagon® when applied to venous leg ulcers in humans, and to obtain further information on the most appropriate dose or doses to apply. A proposed randomised controlled trial aims to further evaluate Nexagon® by randomly allocating (e.g., by the toss of a coin) 90 people with venous leg ulcers to Nexagon® (one of two different doses) or a vehicle (substance containing no medication) to be applied to their ulcer three times over four weeks. Participants will be followed up for 12 weeks to evaluate ulcer healing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of venous leg ulceration
2. Ankle brachial index of > 0.80 measured during screening or within three months prior to the Day -14 visit.
3. Reference ulcer area greater than 1 cm2 and less than 25 cm2
4. Reference ulcer present for at least 4 weeks
5. Have an ankle circumference of greater than 18 cm
6. Male of female patients aged 18 years or over
7. Able to tolerate effective compression bandaging
8. Patients able to walk independently with or without mobility aids
9. Able and willing to give informed consent
10. Able and willing to attend all follow up visits

Exclusion Criteria:

1. Significant change in ulcer size in the screening period screening period
2. Presence of a non-study ulcer within 2.0 cm of the reference ulcer
3. Wound bed with exposed bone, tendon or fascia
4. Patients with leg ulceration etiology other than venous insufficiency
5. Patients who require wheel chairs for normal mobility
6. Patients who have any ulcer (reference or non-reference) which shows signs of clinical infection
7. Patients who have any ulcer (reference or non-reference) positive for β-hemolytic streptococcus upon culture.
8. Patients who are unable to tolerate or comply with the standardized compression bandaging protocol specified in this protocol
9. Female patients who are pregnant or breastfeeding.
10. Patients who are currently taking:

    1. Pentoxifylline (Trental®)
    2. Immunosuppressive therapy
    3. Oral corticosteroid therapy or topical corticosteroid on the leg where the reference ulcer is located
    4. Growth factors (e.g. Regranex)
    5. Cell cultures or topical skin factors
11. Patients with:

    1. Renal insufficiency defined as an estimated GFR which is < 30 mL/min/1.7m2
    2. Abnormal blood biochemistry defined as 3 times that of the upper limit of the normal range
    3. Hepatic insufficiency defined as total bilirubin > 2 mg/dL or serum albumin < 25 g/L
    4. HbA1c > 8.5%
    5. Hemoglobin < 10 g/dL
    6. Hematocrit < 0.30
    7. Platelet count < 100,000
12. Patients have had a myocardial infarction within the previous 6 months or patients with unstable angina pectoris
13. Patients with:

    1. Collagen vascular disease
    2. Severe rheumatoid arthritis
    3. Cellulitis or osteomyelitis
14. Patients who have, or are suspected of having malignancy, or who have received treatment for any active malignancy, apart from non-melanomatic skin cancer, within 3 months prior to treatment
15. Patients who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study, e.g., known to abuse alcohol or drugs currently or to have psychological disorders that could affect follow-up care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rate of reduction in the size of the reference ulcer from Day 0 to Day 28 as measured by photographic planimetry

SECONDARY OUTCOMES:
Complete healing of the treated Venous Leg Ulcer
Reference ulcer wound healing as assessed by digital photographic planimetry
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Scott Bannan, Study Director — OcuNexus Therapeutics, Inc.
Locations (10):
- United States (4):
  - Centre for Clinical Research, San Francisco, California
  - Pacific Wound Center, Stockton, California
  - Penn North Centers for Advanced Wound Care, Erie, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
- New Zealand (6):
  - Waitemata District Health Board, Auckland, Auckland
  - District Nursing and Leg Ulcer Service A+Links Home Health, Auckland
  - Home Health Services Papakura, Auckland
  - Nurse Maude, Christchurch
  - Dunedin Hosptial, Dunedin
  - Waikato Hospital, Hamilton